CLINICAL TRIAL: NCT00858078
Title: A Qualitative Exploration of the Impact of Positive BRCA 1/2 Mutation Status on the Lives of Young Women
Brief Title: A Qualitative Exploration of the Impact of Positive BRCA1/2 Mutation Status on the Lives of Young Women
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909074; 09-C-N074; NCT00954239 (obsolete NCT alias)
Record Dates: First submitted 2009-03-06; First posted 2009-03-09 (Estimated); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: BRCA1 Gene; BRCA2 Gene
Keywords: Qualitative Research; Semi-Structured Telephone Interview; BRCA 1/2; Psychosocial/Behavioral Research; Hereditary Cancer Risk
MeSH Terms: conditions — Fanconi Anemia, Complementation Group D1

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other

GROUPS / COHORTS (2):
- Previously referred: Previously-enrolled subjects from NCI Protocol 01-C-0009
- Self-referred: Self-referred women at increased familial risk of breast and ovarian cancer were recruited through an hereditary breast/ovarian cancer advocacy group

SUMMARY:
Background:

* Mutations detected in the BRCA1 or BRCA2 genes have been show to produce very high risks of breast and ovarian cancer (as high as 90% and 60%, respectively), as well as accompanying risks for several other types of cancer. Women who have these genetic anomalies and who do not have cancer are aware of their high-risk status, which can have an effect on their ability to make decisions about personal choices and health care.
* Researchers are interested in learning more about how people who know their cancer risk status make decisions on personal relationships, family formation, and risk-reduction options.

Objectives:

- To study young women s experiences and decision-making processes regarding family history, genetic testing, couple relationships, family formation, and cancer risk management within the context of their experiences as BRCA1/2 mutation carriers.

Eligibility:

* Women between the ages of 18 and 35 years of age and older who have been identified as having a BRCA1 or BRCA2 mutation. Participants must be contemplating or have experienced couple relationships, family formation, and/or risk management and reduction.
* Participants must be willing to have their interviews digitally recorded

Design:

* Researchers will conduct between 30 and 50 telephone interviews of study participants. Each interview will be approximately 90 minutes in length. The interview consists of open-ended questions that ask about the participants and their experiences before, during, and after they underwent genetic testing for BRCA1/2.
* At least one focus group will be coordinated at a national conference for individuals who are aware of their genetically based cancer risk. If more than 25 individuals are interested in participating in the group, an additional focus group will be convened.
* No medical treatments are specifically offered as a part of this study.

DETAILED DESCRIPTION:
Background:

* BRCA1/2 mutations are present in approximately 1 in 800 individuals in the US, with higher frequency among some populations (e.g., Ashkenazi Jews)
* Mutations confer a lifetime breast cancer risk approaching 90%, ovarian cancer risk as high as 60%, and lesser increases in absolute risks of selected other cancers (e.g., male breast, prostate, pancreas).
* We have successfully conducted follow-up interviews with women in our original studies who had known about their mutations for less than six months, and have gleaned useful longitudinal data. We now propose to conduct additional follow-up interviews with participants who were in the process of making significant decisions about risk-management, relationships, family formation, and other pertinent issues at the time of their initial interviews.
* Additionally, previous research indicates that women who undergo genetic testing very early in young adulthood (i.e., prior to their 25th birthdays) have genetic counseling and support needs that are different from the broader BRCA-positive population.
* Research regarding how these very young mutation carriers manage and accommodate their risk is scarce. We propose to conduct two focus groups with women who considered and/or underwent genetic testing for BRCA prior to their 25th birthdays, who are attending the Joining FORCES annual conference in Orlando, FL June 23-25, 2011.
* The Study Application has been updated with this amendment to reflect the following changes: 1) the inclusion of males who may be enrolled only in the Family Group Interview component of the study & 2) the inclusion older individuals as some women may wish to include male or older members of their family in Family Group Interview portion of the study. To reflect this change the maximum age for study participants has been increased to 100 years of age and males are no longer listed as excluded from the study.

Objectives:

* For follow-up to previous study:

  -- Conduct follow-up telephone interviews with participants who were newly-tested at the time of original data collection to increase understanding of their mutation-positive experience longitudinally.
* For 25 & Under study:

  * Conduct two (2) focus group sessions at the Joining FORCES Annual Conference, focusing on the unique genetic counseling and support needs of women who consider or undergo genetic testing for BRCA1/2 prior to age 25.

Eligibility:

* For follow-up to previous study:

  -- Individuals who were in the process of making decisions relative to their status as mutation positive at the time of their previous interviews will be re-interviewed, in order to learn about their longitudinal experiences and expand the data set.
* For 25 & Under study:

  * Women aged 18-24 who have received a positive BRCA1/2 mutation test result.
  * Women aged 25-30 who considered or completed genetic testing for BRCA1/2 prior to their 25th birthdays
  * English-speaking
  * Attending the 2011 Joining FORCES Annual Conference.

Design:

* For follow-up to previous study:

  * Individuals will be invited to participate in a second telephone interview, during which they will be asked to describe their mutation-related experience since their previous interviews (approximately two years ago).
  * Questions for each participant will be specifically tailored based on their previous interview data. Telephone interviews are anticipated to be approximately 60 minutes in length.
  * **Note: In cases where an individual eligible for follow-up is also participating in the multi-generational family interview (see Amendment A), the individual interview conducted as part of that study will take the place of a follow-up telephone interview.
* For 25 & Under Study

  * Individuals who meet eligibility criteria will be invited to participate in either of two focus group sessions being held during the FORCE conference.
  * Following the conference, each participant will be contacted via telephone to complete a brief family history interview, in order to provide context for the data collected during the focus group.
  * Focus groups will be conducted using a prepared guide (see attachment).
  * Participants will be entered into a raffle at each session, and one participant in each session will win a $50 gift card.
  * Focus group sessions and telephone family history interviews will be audio recorded; then, they will be transcribed and analyzed using modified grounded theoretical design and QSR NVivo v8 software.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must be biologically female
* Participants must have reached their 18th birthday but not have passed their 35th birthday
* Participants must be able to speak and understand English with a level of fluency sufficient for completion of the recorded telephone interview
* Participants must have completed genetic testing for BRCA1/2 and received a positive test result (i.e., a deleterious or disease-related mutation was identified).
* Participants must have experienced or be contemplating/planning couple relationship(s), formation of a family, and/or utilization of risk management/reduction strategies at some point.

EXCLUSION CRITERIA:

-Potential participants will be excluded from the study if they do not agree to have their interview or focus group contributions audio recorded.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Young BRCA1/2 mutation carriers who meet the study criteria.@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2011-06-21 (Actual); Primary Completion 2015-03-13 (Actual); Study Completion 2015-04-03 (Actual)

PRIMARY OUTCOMES:
Telephone Interviews | ongoing
  Conduct follow-up telephone interviews with participantswho were newly-tested at the time of original data collection to increase understanding of their mutationpositive experience longitudinally.
Focus Group Sessions | ongoing
  Conduct two (2) focus group sessions at the JoiningFORCES Annual Conference, focusing on the unique geneticcounseling and support needs of women who consider or undergo genetic testing for BRCA1/2 prior to age 25.

CONTACTS AND LOCATIONS:
Overall Officials: Payal P Khincha, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Werner-Lin A, Hoskins LM, Doyle MH, Greene MH. 'Cancer doesn't have an age': genetic testing and cancer risk management in BRCA1/2 mutation-positive women aged 18-24. Health (London). 2012 Nov;16(6):636-54. doi: 10.1177/1363459312442420. Epub 2012 Apr 30. PMID 22547552
- [Background] Hoskins LM, Roy KM, Greene MH. Toward a new understanding of risk perception among young female BRCA1/2 "previvors". Fam Syst Health. 2012 Mar;30(1):32-46. doi: 10.1037/a0027276. PMID 22429077
- [Background] Hoskins LM, Greene MH. Anticipatory loss and early mastectomy for young female BRCA1/2 mutation carriers. Qual Health Res. 2012 Dec;22(12):1633-46. doi: 10.1177/1049732312458182. Epub 2012 Aug 27. PMID 22927701